CLINICAL TRIAL: NCT02262936
Title: A Randomized Double-blinded Trial Comparing DEsmopressin to FEsoterodine in the Treatment of Severe Nocturia in Women Aged 65 and olDer: The DEFEND Trial
Brief Title: Comparison Between Desmopressin and Fesoterodine for Treatment of Night Time Voiding in Women Aged 65 and Older
Acronym: DEFEND
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Poor recruitment
Sponsor: Mount Sinai Hospital, Canada (Other)
Collaborators: Baycrest (Other); The Physicians' Services Incorporated Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 14-0188-A; 14-56 (Other: Baycrest); 14-16 (Other Grant/Funding Number: Physician Services' Incorporated Foundation)
Record Dates: First submitted 2014-10-08; First posted 2014-10-13 (Estimated); Last update posted 2016-11-15 (Estimated); Status verified 2016-11

CONDITIONS: Nocturia
Keywords: Aged; Deamino Arginine Vasopressin; Fesoterodine; Randomized Controlled Trial
MeSH Terms: conditions — Nocturia | interventions — Deamino Arginine Vasopressin; fesoterodine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Desmopressin (Active Comparator): Patients randomized to receive Desmopressin will be given 0.1mg daily by mouth at bedtime. After 4 weeks, patients will have the option to increase their dose to 0.2mg daily by mouth at bedtime. Total time of drug administration will be 12 weeks.
  Interventions: Drug: Desmopressin
- Fesoterodine (Active Comparator): Patients randomized to receive Fesoterodine will be given 4mg daily by mouth at bedtime. After 4 weeks, patients will have the option to increase their dose to 8mg daily by mouth at bedtime. Total time of drug administration will be 12 weeks.
  Interventions: Drug: Fesoterodine

INTERVENTIONS:
Drug: Desmopressin
  Arms: Desmopressin
Drug: Fesoterodine
  Arms: Fesoterodine

SUMMARY:
Nocturia, or voiding at night, is an extremely troublesome symptom which is highly prevalent in the elderly. Desmopressin is a treatment for nocturia but it can result in hyponatremia (low blood sodium), particularly in those aged 65 and older. Fesoterodine is used for the treatment of overactive bladder (OAB). Recent trials showed Fesoterodine was effective in reducing nocturia. This study aims to answer the following: In women 65 and older with severe nocturia, is Fesoterodine more effective than Desmopressin in reducing the number of night time voids? Does Fesoterodine have a better side effect profile compared to Desmopressin?

The study design is a 12 week randomized double-blinded trial of Fesoterodine and Desmopressin in the treatment of severe nocturia in women aged 65 and older. This will be conducted at the Urogynecology Unit at Mount Sinai Hospital (MSH) and Baycrest. A 3 day voiding diary and Nocturia, Nocturnal Enuresis and Sleep-interruption Questionnaire (NNES-Q) will be completed at baseline and at week 12. The primary outcome will be the number of night time voids in the Fesoterodine group compared to the Desmopressin group, 12 weeks after starting treatment. Secondary outcomes include changes in the NNES-Q scores and the safety of each medication.

This study is expected to show that, in women 65 and older with severe nocturia, Fesoterodine will be more effective in reducing the number of night time voids, reducing the volume of voided urine, increasing the duration of sleep prior to first nocturnal void and improving quality of life relative to Desmopressin. Fesoterodine will also be better tolerated, with fewer significant adverse events, relative to Desmopressin.

DETAILED DESCRIPTION:
This study will include female patients 65 years and older from the Urogynecology Units at Mount Sinai Hospital (MSH) and Baycrest. It will be a 12 week prospective, randomized double-blind trial comparing treatment of nocturia using Fesoterodine and Desmopressin. Patients who agree to participate in the study will receive a starting dose of either Fesoterodine 4mg tablet at bedtime or Desmopressin 0.1mg tablet at bedtime. After 4 weeks, if patients have had minimal improvement in their symptoms and are not significantly affected by side effects, patients will have the option of increasing the dose of their medication to 8mg of Fesoterodine or 0.2mg of Desmopressin. This decision will be made by the patient and physician together.

Patients will undergo block randomization by pharmacy. All patients and investigators will be blinded to the treatment group. Patients will be followed for 12 weeks, with visits at 4 and 12 weeks. Patients will also have urine cultures and uroflowmetry with measurement of post-void residuals at these visits, as per clinic standard of care. Venipuncture to monitor electrolyte levels will be done at baseline, 1 week after randomization and then monthly until the end of the study. If patients choose to increase their dose at the 4 week visit, electrolyte levels will be repeated one week after the dose adjustment and then monthly until the end of the study. The last follow up is at 12 weeks, when a 3 day voiding diary and the NNES-Q will be collected.

ELIGIBILITY:
Inclusion Criteria:

* Menopausal female patients aged 65 years and older
* Patients with severe nocturia, defined as waking to void 3 or more times at night due to an urge to void
* Patients capable of understanding and having signed the consent form after full discussion of the research, nature of the treatment, its risks and benefits

Exclusion Criteria:

* Urinary tract infection or chronic inflammation such as interstitial cystitis and bladder stones
* Urinary and gastric retention
* Narrow-angle glaucoma
* von Willebrand's disease
* Chronic severe constipation or history of gastrointestinal obstructive disease
* Untreated congestive heart failure and venous insufficiency
* Untreated hypertension or tachycardia
* Untreated renal or liver disease
* Untreated diabetes mellitus or insipidus
* Unexplained and untreated electrolyte disturbances
* Any clinical condition which in the opinion of the investigator would not allow safe completion of the study
* Current use of diuretics with untreated electrolyte disturbances
* Patients taking drugs known to be strong CYP3A4 inhibitors (protease inhibitors, ketoconazole, clarithromycin) or strong CYP3A4 inducers (carbamazepine, phenytoin, St. John's Wort) used on a regular basis
* Patients taking anticholinergic or antispasmodic medications who did not comply with a minimum 14 days washout period
* Previous failed therapy with Fesoterodine or Desmopressin
* Hypersensitivity or intolerance to Fesoterodine or Desmopressin
* Hypersensitivity to soya, peanuts or lactose
* Clinically significant outlet obstruction as determined by the investigator
* Patients with Post Void Residual (PVR) > 100 ml
* Patients with Mini-Mental State Exam (MMSE) <24

Min Age: 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 4 (Actual)
Dates: Start 2015-07; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Number of night time voids | 18 months
  Patients will complete a 3-day voiding diary at baseline and after 12 weeks of treatment. The number of night time voids will be compared before and after treatment. The anticipated reduction in night time voids between the two treatment groups will be compared.

SECONDARY OUTCOMES:
Adverse event profile | 18 months
  Type and number of adverse events will be collected and compared between the two treatment groups.
Quality of life | 18 months
  Quality of life, as measured by the Nocturia, Nocturnal Enuresis and Sleep-interruptions Questionnaire (NNES-Q) will be compared between the two treatment groups.
Nocturnal voided volume | 18 months
  The total volume of urine voided at night will be compared between the two treatment groups.
Time to first nocturnal void | 18 months
  The number of minutes of sleep prior to first waking at night to void will be compared between the two treatment groups.

CONTACTS AND LOCATIONS:
Overall Officials: Harold P Drutz, MD, Principal Investigator — MOUNT SINAI HOSPITAL
Locations (1):
- Mount Sinai Hospital, Toronto, Ontario, Canada